CLINICAL TRIAL: NCT02128659
Title: Sexual Health Empowerment for Cervical Health Literacy and Cancer Prevention
Acronym: SHE Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Megha Ramaswamy, PhD, MPH (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Megha Ramaswamy, PhD, MPH, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13559; R01CA181047-01A1 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHE Project (Experimental): Receives SHE Project Intervention during Week 1 of enrollment
  Interventions: Behavioral: SHE Project
- Wait-List Control (Active Comparator): Receive SHE Project intervention during Week 2 of Enrollment
  Interventions: Behavioral: SHE Project

INTERVENTIONS:
Behavioral: SHE Project — Consists of five-sessions, starting on a Monday and ending Friday. Each day involves an approximately 2 hour session.

SUMMARY:
The purpose of this study is to learn if a cervical health literacy program is a practical and helpful way of improving women's cervical health knowledge and improving cancer screening behaviors, and ultimately preventing cervical cancer.

DETAILED DESCRIPTION:
Women in the criminal just system are 4-5 times more likely to have cervical cancer than non-incarcerated women. Little is known about how to close this gap. The few investigators that have studied cervical cancer risk and disease among women in jails and prisons have found that while many women get screened for cervical cancer, less than half get follow-up care.

The investigator's pilot research suggests the most important contributor to cervical cancer risk, and perhaps lack of follow-up, is incarcerated women's low health literacy about both cervical cancer and broader reproductive health issues. This study is testing a sexual health empowerment intervention (SHE Project) to see if it improves incarcerated women's reproductive health literacy.

ELIGIBILITY:
Inclusion Criteria:

* Women sentenced or anticipate a sentence of one year or less
* Ability to follow participants post-jail release
* Able to read and understand English

Exclusion Criteria:

* Women who have been treated for cervical cancer with procedures that would obviate the need for regular screening
* Exhibit severe psychological distress

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of sexual health empowerment (SHE Project) intervention | Change from Baseline to 5 days
  Changes in knowledge, beliefs, and self-efficacy pre- and post-intervention measured using data collection instruments (Pap Knowledge Scale, Health Belief Model Scale for Cervical Cancer and Pap Smear Test, Self-Efficacy Scale for Pap Smear Screening Participation, Investigator developed study specific survey specific to women with criminal justice involvement, 10-question satisfaction survey)

SECONDARY OUTCOMES:
Long-term health behavior | 6 Months post-jail release
  Participant screening behaviors (Paps or Sexually Transmitted Infections [STIs]), clinical follow-up of screening, and strategies for navigating health care encounters. Measured using self-report of screening and clinical follow-up survey, review of participant medical charts)
Long-term health behavior | 12 Months post-jail release
  Participant screening behaviors (Paps or STIs), clinical follow-up of screening, and strategies for navigating health care encounters. Measured using self-report of screening and clinical follow-up survey, review of participant medical charts)
Long-term health behavior | 24 Months post-jail release
  Participant screening behaviors (Paps or STIs), clinical follow-up of screening, and strategies for navigating health care encounters. Measured using self-report of screening and clinical follow-up survey, review of participant medical charts)
Long-term health behavior | 36 months post-jail release
  Participant screening behaviors (Paps or STIs), clinical follow-up of screening, and strategies for navigating health care encounters. Measured using self-report of screening and clinical follow-up survey, review of participant medical charts)

CONTACTS AND LOCATIONS:
Overall Officials: Megha Ramaswamy, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - Wyandotte County Detention Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Jackson County Detention/Regional Correctional Center, Kansas City, Missouri

REFERENCES:
- [Background] Pickett ML, Allison M, Twist K, Klemp JR, Ramaswamy M. Breast Cancer Risk Among Women in Jail. Biores Open Access. 2018 Sep 20;7(1):139-144. doi: 10.1089/biores.2018.0018. eCollection 2018. PMID 30250761
- [Background] Kelly PJ, Emerson A, Fair C, Ramaswamy M. Assessing fidelity: balancing methodology and reality in jail interventions. BMC Womens Health. 2018 Jul 23;18(1):127. doi: 10.1186/s12905-018-0617-x. PMID 30037333
- [Background] Emerson AM. Narrative Inquiry Into Shelter-Seeking by Women With a History of Repeated Incarceration: Research and Nursing Practice Implications. ANS Adv Nurs Sci. 2018 Jul/Sep;41(3):260-274. doi: 10.1097/ANS.0000000000000216. PMID 29901467
- [Background] Emerson AM. Strategizing and Fatalizing: Self and Other in the Trauma Narratives of Justice-Involved Women. Qual Health Res. 2018 May;28(6):873-887. doi: 10.1177/1049732318758634. Epub 2018 Feb 24. PMID 29478403
- [Background] Kelly PJ, Ramaswamy M. Closing the cervical cancer disparity gap. Public Health Nurs. 2017 May;34(3):195-196. doi: 10.1111/phn.12336. No abstract available. PMID 28493356
- [Background] Ramaswamy M, Lee J, Wickliffe J, Allison M, Emerson A, Kelly PJ. Impact of a brief intervention on cervical health literacy: A waitlist control study with jailed women. Prev Med Rep. 2017 Apr 5;6:314-321. doi: 10.1016/j.pmedr.2017.04.003. eCollection 2017 Jun. PMID 28435785
- [Background] Kelly PJ, Hunter J, Daily EB, Ramaswamy M. Challenges to Pap Smear Follow-up among Women in the Criminal Justice System. J Community Health. 2017 Feb;42(1):15-20. doi: 10.1007/s10900-016-0225-3. PMID 27449030
- [Background] Ramaswamy M, Kelly PJ. "The Vagina is a Very Tricky Little Thing Down There": Cervical Health Literacy among Incarcerated Women. J Health Care Poor Underserved. 2015 Nov;26(4):1265-85. doi: 10.1353/hpu.2015.0130. PMID 26548678
- [Background] Ramaswamy M, Simmons R, Kelly PJ. The development of a brief jail-based cervical health promotion intervention. Health Promot Pract. 2015 May;16(3):432-42. doi: 10.1177/1524839914541658. Epub 2014 Jul 25. PMID 25063589